CLINICAL TRIAL: NCT04318600
Title: Allogeneic Amniotic Mesenchymal Stem Cell Therapy for Lupus Nephritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Collaborators: The First People's Hospital of Yunnan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014001
Record Dates: First submitted 2020-03-11; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2014-01

CONDITIONS: Lupus Nephritis; Mesenchymal Stem Cells
Keywords: Lupus Nephritis; Human Amniotic Mesenchymal Stem Cell; cell therapy; clinical trail
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- human amniotic mesenchymal stem cell treatment group (Experimental)
  Interventions: Drug: human amniotic mesenchymal stem cell
- blank control group (No Intervention)

INTERVENTIONS:
Drug: human amniotic mesenchymal stem cell — human amniotic mesenchymal stem cell (hA-MSC) for the treatment of lupus nephritis patients with WHO class III, IV or V LN were given hA-MSC (Peripheral intravenous infusion, dose 1×106/kg cells, once every month for three times).
  Arms: human amniotic mesenchymal stem cell treatment group

SUMMARY:
This study would further evaluate the safety and efficacy of human amniotic mesenchymal stem cell (hA-MSC) for the treatment of lupus nephritis (LN).

DETAILED DESCRIPTION:
Eleven patients with WHO class III, IV or V LN were given hA-MSC (Peripheral intravenous infusion, dose 1×106/kg cells, once every month for three times). At the same time, five patients with LN who were not given hA-MSC as the blank control group. All patients did not received intravenous corticosteroids pulse therapy, but the use of oral corticosteroids and intravenous cyclophosphamide, or oral mycophenolate mofetil, tacrolimus , leflunomide were allowed.

ELIGIBILITY:
Enrollment criteria:

* Adult patients (age 14-60 years) who were diagnosed as lupus nephritis, regardless of gender, uncontrolled disease course;
* Pathological examination of puncture biopsy resulting in diagnosis of type II, III, or IV lupus nephritis;
* SLEDAI score >8;
* proteinuria greater than 1 g/day and active urinary sediments;
* Lupus nephritis treatment according to guidelines and norms before human amniotic mesenchymal stem cells therapy;
* If there is a possibility of pregnancy in female, must be negative pregnancy test, not in lactation, and confirm that is receiving the method of contraception recognized by the researchers, and agree to maintain the method of contraception throughout the study. Sexually active male patients must agree to the use of an appropriate contraceptive method for birth control from the first administration of the study treatment until 24 weeks after the last administration.
* The subjects should be fully informed, voluntarily sign the informed consent, and agree to participate in all visits, examinations, and treatments as required by the experimental protocol.

Exclusion criteria:

* Patients with kidney biopsy diagnosis of type I, VI lupus nephritis or a diagnosis of another glomerular disease;
* Patients with abnormal renal function (serum creatinine ≥ the upper limit of normal);
* Patients with active liver disease or abnormal liver function test results (ALT or AST ≥2 times the upper limit of normal);
* Patients with blood leukocyte count <2.5 × 109/L, hemoglobin <90 g/L, platelet count <100 × 109/L, or those who have other hematologic diseases (severe anemia, idiopathic thrombocytopenic purpura, splenomegaly, coagulation dysfunction, etc.);
* Patients with serious and unstable cardiovascular or cerebrovascular diseases (unstable angina pectoris, coronary artery disease, cerebrovascular disease, transient ischemic attack, congestive heart failure, etc.), acute and difficult to control the disease, after treatment has not been effectively controlled severe hypertension (blood pressure >160/100 mm Hg), or organ transplantation;
* Patients with uncontrolled infection;
* Patients with tumors or abnormal tumor marker levels; 8. Patients with blood-borne diseases (i.e., HIV, syphilis, hepatitis B, and hepatitis C);
* Pregnancy, the potential for pregnancy, or lactation;
* Patients with a history of allergy, especially patients allergic to human blood albumin;
* Patients with mental illness affecting their voluntarism, ability to make decisions, and ability to communicate；
* A history of alcoholism or known drug addiction in the last 2 years;
* Participation in another clinical trial within the last 3 months;
* Patients judged inappropriate for this study by the physicians.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 60 weeks
  The patient's discomfort and clinical symptoms during the study were recorded, as well as the related laboratory test indicators and physical examination abnormalities of the subjects during the study. Describe the association with Amniotic mesenchymal stem cell therapy and calculate the incidence of treatment-related acute and chronic adverse events.

SECONDARY OUTCOMES:
Changes in 24h urine protein quantification before and after treatment； | 60 weeks
  24-hour urinary protein quantification from baseline to 60 weeks of treatment.
Changes in eGFR before and after treatment; | 60 weeks
  changes in estimated glomerular filtration rate (eGFR) from baseline to 60 weeks of treatment.
Changes in SLEDAI score before and after treatment； | 60 weeks
  changes in SLEDAI score from baseline to 60 weeks of treatment. SLEDAI score: 0~4 points basically no activity;5-9 minutes light activity;10-14 minutes of moderate activity;≥15 minutes of severe activity.

REFERENCES:
- [Derived] Naeem A, Gupta N, Naeem U, Khan MJ, Elrayess MA, Cui W, Albanese C. A comparison of isolation and culture protocols for human amniotic mesenchymal stem cells. Cell Cycle. 2022 Aug;21(15):1543-1556. doi: 10.1080/15384101.2022.2060641. Epub 2022 Apr 12. PMID 35412950